CLINICAL TRIAL: NCT01313000
Title: Pilot Study To Evaluate Upper Arm Autologous Fat Transfer
Brief Title: Study To Evaluate Upper Arm Autologous Fat Transfer
Status: Completed | Type: Observational
Sponsor: Sound Surgical Technologies, LLC. (Industry)
Responsible Party: David Matlock, Vaser HiDef Liposculpturing Institute of Beverly Hills
Other Study IDs: SST2001-1
Record Dates: First submitted 2011-03-09; First posted 2011-03-11 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2012-03

CONDITIONS: Cosmetic and Circumferential Change After Fat Transfer
Keywords: fat, transfer, autologous fat transfer, bicep
MeSH Terms: conditions — Platelet Glycoprotein IV Deficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Autologous fat transfer
  Interventions: Procedure: Autologous fat transfer

INTERVENTIONS:
Procedure: Autologous fat transfer — Autologous fat transfer from abdomen to upper arms

SUMMARY:
The objective of this pilot study is to observe the utility of autologous transfer of fat collected using ultrasonic assisted liposuction into the upper arms with ultrasonic visualization.

ELIGIBILITY:
Inclusion Criteria:

1. Is male.
2. Is between 20 and 50 years of age, inclusive, on the day of enrolment.
3. Is to undergo abdominal liposuction.
4. Wishes to undergo autologous fat transfer to the upper arms.

Exclusion Criteria:

1. Currently enrolled in another device or drug study that has not completed the required follow-up period, or has completed all other study-required follow-up less than 30 days before enrolment in this study.
2. Undergoing body contouring for reconstruction following injury or disease.
3. Deemed inappropriate candidates for the surgical procedures for any reason.
4. Are unwilling to undergo the study procedures or participate fully in all follow-up.

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Male patients undergoing abdominal liposuction who wish autologous fat transfer to the upper arms
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2011-03; Primary Completion 2011-12 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Dr David Matlock, Beverly Hills, California, United States